CLINICAL TRIAL: NCT00189423
Title: ResQ Trial: Comparison of Standard CPR Alone Versus Active Compression Decompression CPR Plus an ITD on Survival From Out-of-Hospital Cardiac Arrest
Brief Title: ResQ Trial: Impact of an ITD and Active Compression Decompression CPR on Survival From Out-of-Hospital Cardiac Arrest
Acronym: ResQ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of funding. Follow-up completed for all enrolled subjects.
Sponsor: Advanced Circulatory Systems (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 265; R44HL065851-03 (NIH); 2R44HL065851-03 (NIH); 43-0303-000; NCT00225953 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Heart Arrest; Death, Sudden, Cardiac; Cardiopulmonary Resuscitation; Cardiac Arrest
Keywords: Heart Arrest; Cardiac Arrest; Cardiopulmonary Resuscitation; Impedance Threshold Device; Active Compression Decompression; ResQPOD; ResQPump; Survival; Out-of-hospital; Prehospital; ResQCPR System
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active compression decompression cardiopulmonary resuscitation (ACD-CPR) with an impedance threshold device (ITD)
  Interventions: Device: Use of an impedance threshold device (ITD) during the performance of active compression decompression CPR (ACD-CPR)
- 2 (Active Comparator): Conventional standard cardiopulmonary resuscitation (S-CPR)
  Interventions: Procedure: Standard cardiopulmonary resuscitation (S-CPR)

INTERVENTIONS:
Device: Use of an impedance threshold device (ITD) during the performance of active compression decompression CPR (ACD-CPR) — The ITD selectively prevents the influx of unnecessary respiratory gases into the patient during the chest wall recoil phase of CPR.
  The ResQPump, a hand-held device containing a suction cup, attaches to the chest and actively compresses and actively re-expands the chest during the performance of CPR.
  Other Names: Impedance threshold device: ResQPOD CE CA; Device used to perform ACD-CPR: ResQPump
  Arms: 1
Procedure: Standard cardiopulmonary resuscitation (S-CPR) — Conventional standard cardiopulmonary resuscitation (S-CPR)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether performing active compression decompression cardiopulmonary resuscitation (ACD-CPR) with an impedance threshold device (ITD) compared to conventional standard cardiopulmonary resuscitation (S-CPR) will impact the neurologic recovery and survival to hospital discharge following out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
Despite receiving conventional, standard CPR (S-CPR), most patients who experience out-of-hospital cardiac arrest die prior to arriving at a hospital. At the present time, the hospital discharge rate following out-of-hospital, nontraumatic cardiac arrest in adults in the United States is estimated to be less than 5%. Many factors contribute to the current poor survival statistics, including the inefficiency of the technique itself. CPR provides only 10% to 20% of normal myocardial perfusion, and only 20% to 30% of physiologically normal cerebral perfusion.

A new method of CPR that combines ACD and an ITD (ACD-CPR+ITD) has been shown in animal models and in clinical trials conducted in Europe to provide significantly more blood flow to the vital organs and to improve survival rates when compared to S-CPR or ACD-CPR alone.

ACD-CPR+ITD works by decreasing intrathoracic pressure during the chest wall recoil (or decompression) phase of CPR, creating a vacuum within the thorax relative to the rest of the body. When compared with controls, use of ACD-CPR+ITD (a) enhances blood return to the thorax during the chest wall recoil phase, (b) enhances blood flow to the heart and brain, (c) provides real-time feedback to rescuers to maintain high-quality CPR, (d) improves overall CPR efficiency and, as a result of the forgoing, (e) improves short-term survival rates.

The sponsor and others recently evaluated the effectiveness of the combination of conventional, manual standard CPR±ITD in animals and humans. The ITD increased short-term survival rates in these studies as well. Two clinical trials were performed in Milwaukee, Wisconsin, under IDE (#G980125). Both compared S-CPR with either a sham (nonfunctional or placebo) or active (functional) ITD. The results from the hemodynamic study demonstrated that systolic blood pressure, the primary end point, increased from approximately 45 mmHg with the sham ITD to approximately 85 mmHg with the active ITD (P less than 0.05). Intensive care unit admission rate was the primary end point of the clinical outcome study.

Comparisons: The objective of this two-arm, multisite, randomized, pivotal IDE clinical trial is to compare survival to hospital discharge with neurologic recovery rates in subjects receiving S-CPR compared to ACD-CPR+ITD following out-of-hospital cardiac arrest in well-established American emergency medical services systems.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects initially presumed or known to be 18 years of age or older
* Subjects who present with out-of-hospital cardiac arrest from presumed cardiac etiology and who receive CPR by Emergency Medical Services (EMS) personnel for at least 1 minute
* Subjects whose airways are managed with a cuffed ET tube, combitube, or laryngeal mask airway or facemask

Exclusion Criteria:

* Adult subjects presumed or known to be less than 18 years of age
* Subjects with known or likely traumatic injuries causing cardiac arrest or cardiac arrest of presumed noncardiac origin
* Subjects with preexisting Do Not Resuscitate (DNR) orders
* Subjects with signs of obvious clinical death or conditions that preclude the use of CPR
* Family or legal representative request that the subject not be entered into the study
* Subjects experiencing in-hospital cardiac arrest
* Subjects with a recent sternotomy with wound not appearing completely healed (if unknown) or less than 6 months (if known)
* Subjects who received less than 1 minute of CPR by EMS personnel
* Subjects with a complete airway obstruction that cannot be cleared or in whom attempts at advanced airway management are unsuccessful
* Subjects intubated with a leaky or uncuffed advanced airway device or presence of stomas, tracheotomies, or tracheostomies
* Subjects who rearrest and are encountered by EMS within 365 days of the index cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1653 (Actual)
Dates: Start 2005-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith G. Lurie, MD, Principal Investigator — Advanced Circulatory Systems
Locations (7):
- United States (7):
  - Site 07: Indianapolis, IN, Indianapolis, Indiana
  - Site 06: Washtenaw & Livingston Counties, MI, Ann Arbor, Michigan
  - Site 04: Oakland & Macomb Counties, MI, Royal Oak, Michigan
  - Site 02: Minneapolis, MN, Minneapolis, Minnesota
  - Site 01: St. Paul, MN, Saint Paul, Minnesota
  - Site 03: Whatcom County, WA, Bellingham, Washington
  - Site 05: Oshkosh, WI, Oshkosh, Wisconsin

REFERENCES:
- [Background] Wolcke BB, Mauer DK, Schoefmann MF, Teichmann H, Provo TA, Lindner KH, Dick WF, Aeppli D, Lurie KG. Comparison of standard cardiopulmonary resuscitation versus the combination of active compression-decompression cardiopulmonary resuscitation and an inspiratory impedance threshold device for out-of-hospital cardiac arrest. Circulation. 2003 Nov 4;108(18):2201-5. doi: 10.1161/01.CIR.0000095787.99180.B5. Epub 2003 Oct 20. PMID 14568898
- [Background] Plaisance P, Adnet F, Vicaut E, Hennequin B, Magne P, Prudhomme C, Lambert Y, Cantineau JP, Leopold C, Ferracci C, Gizzi M, Payen D. Benefit of active compression-decompression cardiopulmonary resuscitation as a prehospital advanced cardiac life support. A randomized multicenter study. Circulation. 1997 Feb 18;95(4):955-61. doi: 10.1161/01.cir.95.4.955. PMID 9054757
- [Background] Plaisance P, Soleil C, Lurie KG, Vicaut E, Ducros L, Payen D. Use of an inspiratory impedance threshold device on a facemask and endotracheal tube to reduce intrathoracic pressures during the decompression phase of active compression-decompression cardiopulmonary resuscitation. Crit Care Med. 2005 May;33(5):990-4. doi: 10.1097/01.ccm.0000163235.18990.f6. PMID 15891326
- [Background] Plaisance P, Lurie KG, Vicaut E, Martin D, Gueugniaud PY, Petit JL, Payen D. Evaluation of an impedance threshold device in patients receiving active compression-decompression cardiopulmonary resuscitation for out of hospital cardiac arrest. Resuscitation. 2004 Jun;61(3):265-71. doi: 10.1016/j.resuscitation.2004.01.032. PMID 15172704
- [Background] Voelckel WG, Lurie KG, Zielinski T, McKnite S, Plaisance P, Wenzel V, Lindner KH. The effects of positive end-expiratory pressure during active compression decompression cardiopulmonary resuscitation with the inspiratory threshold valve. Anesth Analg. 2001 Apr;92(4):967-74. doi: 10.1097/00000539-200104000-00032. PMID 11273935
- [Background] Plaisance P, Lurie KG, Vicaut E, Adnet F, Petit JL, Epain D, Ecollan P, Gruat R, Cavagna P, Biens J, Payen D. A comparison of standard cardiopulmonary resuscitation and active compression-decompression resuscitation for out-of-hospital cardiac arrest. French Active Compression-Decompression Cardiopulmonary Resuscitation Study Group. N Engl J Med. 1999 Aug 19;341(8):569-75. doi: 10.1056/NEJM199908193410804. PMID 10451462
- [Background] Schneider T, Wik L, Baubin M, Dirks B, Ellinger K, Gisch T, Haghfelt T, Plaisance P, Vandemheen K. Active compression-decompression cardiopulmonary resuscitation--instructor and student manual for teaching and training. Part I: The workshop. Resuscitation. 1996 Oct;32(3):203-6. doi: 10.1016/0300-9572(96)00946-x. PMID 8923582
- [Background] Wik L, Schneider T, Baubin M, Dirks B, Ellinger K, Gisch T, Haghfelt T, Plaisance P, Vandemheen K. Active compression-decompression cardiopulmonary resuscitation--instructor and student manual for teaching and training. Part II: A student and instructor manual. Resuscitation. 1996 Oct;32(3):206-12. doi: 10.1016/0300-9572(96)82051-x. No abstract available. PMID 8923583
- [Background] Lurie K, Voelckel W, Plaisance P, Zielinski T, McKnite S, Kor D, Sugiyama A, Sukhum P. Use of an inspiratory impedance threshold valve during cardiopulmonary resuscitation: a progress report. Resuscitation. 2000 May;44(3):219-30. doi: 10.1016/s0300-9572(00)00160-x. PMID 10825624
- [Background] Plaisance P, Lurie KG, Payen D. Inspiratory impedance during active compression-decompression cardiopulmonary resuscitation: a randomized evaluation in patients in cardiac arrest. Circulation. 2000 Mar 7;101(9):989-94. doi: 10.1161/01.cir.101.9.989. PMID 10704165
- [Background] Mauer DK, Nolan J, Plaisance P, Sitter H, Benoit H, Stiell IG, Sofianos E, Keiding N, Lurie KG. Effect of active compression-decompression resuscitation (ACD-CPR) on survival: a combined analysis using individual patient data. Resuscitation. 1999 Aug;41(3):249-56. doi: 10.1016/s0300-9572(99)00073-8. PMID 10507710
- [Background] Pirrallo RG, Aufderheide TP, Provo TA, Lurie KG. Effect of an inspiratory impedance threshold device on hemodynamics during conventional manual cardiopulmonary resuscitation. Resuscitation. 2005 Jul;66(1):13-20. doi: 10.1016/j.resuscitation.2004.12.027. PMID 15993724
- [Background] Aufderheide TP, Pirrallo RG, Provo TA, Lurie KG. Clinical evaluation of an inspiratory impedance threshold device during standard cardiopulmonary resuscitation in patients with out-of-hospital cardiac arrest. Crit Care Med. 2005 Apr;33(4):734-40. doi: 10.1097/01.ccm.0000155909.09061.12. PMID 15818098
- [Background] Lurie KG, Zielinski T, McKnite S, Aufderheide T, Voelckel W. Use of an inspiratory impedance valve improves neurologically intact survival in a porcine model of ventricular fibrillation. Circulation. 2002 Jan 1;105(1):124-9. doi: 10.1161/hc0102.101391. PMID 11772887
- [Background] Langhelle A, Stromme T, Sunde K, Wik L, Nicolaysen G, Steen PA. Inspiratory impedance threshold valve during CPR. Resuscitation. 2002 Jan;52(1):39-48. doi: 10.1016/s0300-9572(01)00442-7. PMID 11801347
- [Background] Yannopoulos D, Sigurdsson G, McKnite S, Benditt D, Lurie KG. Reducing ventilation frequency combined with an inspiratory impedance device improves CPR efficiency in swine model of cardiac arrest. Resuscitation. 2004 Apr;61(1):75-82. doi: 10.1016/j.resuscitation.2003.12.006. PMID 15081185
- [Background] Raedler C, Voelckel WG, Wenzel V, Bahlmann L, Baumeier W, Schmittinger CA, Herff H, Krismer AC, Lindner KH, Lurie KG. Vasopressor response in a porcine model of hypothermic cardiac arrest is improved with active compression-decompression cardiopulmonary resuscitation using the inspiratory impedance threshold valve. Anesth Analg. 2002 Dec;95(6):1496-502, table of contents. doi: 10.1097/00000539-200212000-00007. PMID 12456407
- [Background] Frascone RJ, Bitz D, Lurie K. Combination of active compression decompression cardiopulmonary resuscitation and the inspiratory impedance threshold device: state of the art. Curr Opin Crit Care. 2004 Jun;10(3):193-201. doi: 10.1097/01.ccx.0000126089.40242.a9. PMID 15166836
- [Background] Lurie KG, Shultz JJ, Callaham ML, Schwab TM, Gisch T, Rector T, Frascone RJ, Long L. Evaluation of active compression-decompression CPR in victims of out-of-hospital cardiac arrest. JAMA. 1994 May 11;271(18):1405-11. PMID 8176802
- [Background] Voelckel WG, Lurie KG, Sweeney M, McKnite S, Zielinski T, Lindstrom P, Peterson C, Wenzel V, Lindner KH. Effects of active compression-decompression cardiopulmonary resuscitation with the inspiratory threshold valve in a young porcine model of cardiac arrest. Pediatr Res. 2002 Apr;51(4):523-7. doi: 10.1203/00006450-200204000-00020. PMID 11919340
- [Result] Aufderheide TP, Frascone RJ, Wayne MA, Mahoney BD, Swor RA, Domeier RM, Olinger ML, Holcomb RG, Tupper DE, Yannopoulos D, Lurie KG. Standard cardiopulmonary resuscitation versus active compression-decompression cardiopulmonary resuscitation with augmentation of negative intrathoracic pressure for out-of-hospital cardiac arrest: a randomised trial. Lancet. 2011 Jan 22;377(9762):301-11. doi: 10.1016/S0140-6736(10)62103-4. PMID 21251705
- See also: Sponsor: Advanced Circulatory Systems, Inc. home page — http://www.advancedcirculatory.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted under a waiver of informed consent for emergency research that was approved by the U.S. Food and Drug Administration and by the Institutional Review Boards at participating study sites. All adults with out-of-hospital cardiac arrest were eligible for the study.
Pre-assignment Details: All sites were required to complete a run-in phase prior to to beginning randomization. A total of 2667 patients (197 run-in, 2470 pivotal) were provisionally enrolled and received randomized CPR treatment. Of these, 1653 pivotal patients met the final selection criteria (non-traumatic arrest due to cardiac cause).
Groups:
- Standard CPR: Conventional standard cardiopulmonary resuscitation (S-CPR)
- ACD CPR Plus ITD: Active compression decompression CPR plus an Impedance Threshold Device
Period: Overall Study
Arm/Group | Standard CPR | ACD CPR Plus ITD
Started | 813 | 840
Completed | 48 | 74
Not Completed | 765 | 766
Not completed — Death | 746 | 747
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Lost to Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard CPR | ACD CPR Plus ITD | Total
Number analyzed (Participants) | 813 | 840 | 1653
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 377 | 369 | 746
  >=65 years | 436 | 470 | 906
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (14.5) | 67.0 (15.2) | 66.9 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 282 | 556
  Male | 539 | 558 | 1097
Region of Enrollment [Number; unit: participants]
  United States | 813 | 840 | 1653

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Survived to Hospital Discharge With Favorable Neurologic Function Defined as MRS Score <=3
Description: favorable neurologic function is defined as modified Rankin Scale (MRS) score <= 3. Modified Rankin Scale measures functional outcome in stroke. It is a scale of 0-5 where 0=no symptoms at all and 5=severe disability: bedridden, incontinent, and requiring constant nursing care and attention.
Time Frame: When the subject is discharged from the hospital; an average of 12 days after cardiac arrest for subjects surviving to hospital discharge
Population: The population was a modified Intent to Treat (mITT) population who received EMS CPR per study protocol after meeting initial inclusion criteria and who were finally included in the final analysis population after meeting final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 47 | 75
Statistical Analysis 1: Comparison: Standard CPR; Test type: Superiority or Other; p = 0.019, Fisher Exact; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.07 to 2.36]

2. Secondary Outcome: Major Adverse Event Rate as Measured by Number of Patients With One or More Adverse Events
Description: Number of patients with one or more major adverse events, through hospital discharge. Major adverse events included: death, rearrest, pulmonary edema, seizure, bleeding requiring intervention, rib/sterna fracture, pneumothorax, hemothorax, cardiac tamponade, cerebral bleeding, aspiration, internal organ injury.
Time Frame: Time from cardiac arrest through hospital discharge (an average of 12 days for subjects surviving to hospital discharge
Population: Population is a modified Intent to Treat (mITT) population consisting of patients who met all initial and final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 766 | 787
Statistical Analysis 1: Comparison: Standard CPR vs ACD CPR Plus ITD; Test type: Non-Inferiority or Equivalence — non-inferiority margin of 5%; p = 0.0001, Fisher Exact test, for non-inferiority — p value is for non-inferiority with a margin of 5% (exact binomial test)
Statistical Analysis 2: Comparison: Standard CPR vs ACD CPR Plus ITD; Test type: Superiority or Other; p = 0.681, Fisher Exact

3. Secondary Outcome: Return of Spontaneous Circulation (ROSC)
Description: Number of subjects who had ROSC, defined as any return of spontaneous circulation for any duration, reported during resuscitation in the field by EMS.
Time Frame: Time of cardiac arrest until discontinuation of efforts
Population: Population was a modified Intent to Treat (mITT) population that consisted of patients who met all initial and final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 324 | 343

4. Secondary Outcome: Survival to Hospital (e.g., Intensive Care Unit) Admission
Description: Number of patients who survived to hospital or ICU admission after being transported to the emergency department (ED) after out-of-hospital cardiac arrest.
Time Frame: Time of hospital admission, up to 1 day after cardiac arrest
Population: Population is a modified Intent to Treat (mITT) population who received EMS CPR per study protocol after meeting initial inclusion criteria and also met final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 216 | 237

5. Secondary Outcome: Survival to 24 Hours
Description: Number of patients who were alive 24 hours after the initial cardiac arrest.
Time Frame: 24 hours following cardiac arrest
Population: Population is a modified Intent to Treat (mITT) population who met ititial inclusion criteria and final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 176 | 197

6. Secondary Outcome: Survival to Hospital Discharge
Time Frame: cardiac arrest to hospital discharge
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 104 | 80

7. Secondary Outcome: Survival to 90 Days
Description: Number of patients who are known to be alive 90 days after the index cardiac arrest.
Time Frame: 90 days following cardiac arrest
Population: Population is a modified Intent to Treat (mITT) population that met initial and final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 58 | 87

8. Secondary Outcome: Survival to 365 Days
Description: Number of patients who are alive 365 days after the index cardiac arrest.
Time Frame: 365 days following cardiac arrest
Population: Population is a modified Intent to Treat (mITT) population who met initial and final inclusion criteria.
Measure: Number; unit: patients
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 813 | 840
patients | 48 | 74
Statistical Analysis 1: Comparison: Standard CPR vs ACD CPR Plus ITD; Test type: Superiority or Other; p = 0.024, Fisher Exact

9. Secondary Outcome: Neurological Recovery at 1 Year [Measured by Cognitive Abilities Screening Instrument (CASI)]
Description: CASI is scored on a scale of 0-100 with 100 being the best score. The instrument evaluates attention, concentration, and short- and long-term memory as well as language and abstraction. The CASI score is a total score and not an aggregate of subscores.
Time Frame: One year after index arrest
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard CPR | ACD CPR Plus ITD
Number analyzed (Participants) | 41 | 30
units on a scale | 93.7 (11.8) | 94.7 (4.4)

ADVERSE EVENTS:
Time Frame: Through hospital discharge, up to 30 days after index arrest.
Description: Only serious adverse events were assessed for this study.
Arm/Group | Standard CPR | ACD CPR Plus ITD
Serious Adverse Events (participants affected / at risk) | 766/813 | 787/840
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard CPR (N=813) | ACD CPR Plus ITD (N=840)
death (General disorders) | 729 (729) | 734 (734)
re-arrest (General disorders) | 161 (161) | 184 (184)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 62 (62) | 93 (93)
seizure (General disorders) | 13 (13) | 11 (11)
bleeding requiring intervention (General disorders) | 3 (3) | 7 (7)
rib/sterna fracture (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 11 (11)
cerebral bleeding (General disorders) | 3 (3) | 2 (2)
internal organ injury (General disorders) | 0 (0) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10)
hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days